CLINICAL TRIAL: NCT05958147
Title: Concentrated Platelet Rich Fibrin (C-PRF) as Adjunct to Non-surgical Periodontal Therapy- a Split Mouth Randomized Clinical Trail
Brief Title: Concentrated Platelet Rich Fibrin (C-PRF) as Adjunct to Non-surgical Periodontal Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KCDSHEC/IP/2023/P7
Record Dates: First submitted 2023-07-14; First posted 2023-07-24 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probing sites with SPR and C-PRF application (Experimental): The test group received the C-PRF as adjunct to sacling and root planing
  Interventions: Biological: C-PRF
- Probing sites with SPR alone (No Intervention)

INTERVENTIONS:
Biological: C-PRF — thorough scaling and root planing is performed followed by withdraw of 5ml of blood from antecubital vein of patient with consent . Following C-PRF protocol of 3000rpm for 8 min centrifugation is performed. 1ml of plasma is drawn from the test tube just above the red blood cell layer and allowed to clot and the formed clot is placed in the periodontal pocket after scaling and root planing
  Other Names: Concentrated platelet rich fibrin
  Arms: Probing sites with SPR and C-PRF application

SUMMARY:
The current study is a prospective randomised split mouth study to evaluate the effect of concentrated Platelet Rich Fibrin as an adjunct to the scaling and root planing

DETAILED DESCRIPTION:
Twelve healthy individuals satisfying the inclusion and exclusion criteria were recruited for the study. A detailed, thorough medical and dental history was obtained and each patient was subjected to comprehensive clinical and radiological examination. All patients were informed about the nature of the study, procedure involved, potential benefits and risks associated with procedure and written informed consent were obtained from all patients.

All the patients underwent scaling and root planing. As it is split mouth study design the test site is treated with Concentrated platelet rich fibrin( C-PRF) and the contralateral site is not treated with C-PRF. Periodotal pack was placed and patient was recalled after 6 weeks for the follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ranging from 18-45 years
2. Contralateral sites with probing depth 5mm-7mm associated with premolar and molar teeth with no furcation involvement
3. No systemic disease
4. Not under any medication which effect the outcome of periodontal therapy

Exclusion Criteria:

1. History of any periodontal therapy within past 6 months
2. Pregnant and lactating mothers
3. Smokers smoking >10 cigarettes per day
4. Patients with blood disorders or platelet count less than 50000 cells/ µL
5. Patients with known systemic disease
6. Non-compliant patients

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-23 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Probing pocket Depth | 6 weeks
  measured using a UNC-15 probe (university of North Carolina-15 periodontal probe- Hu-Friedy, Chicago, IL, USA)
Relative attachment level | 6 weeks
  measured by placing the acrylic stent on the selected teeth using UNC-15 probe (university of North Carolina-15 periodontal probe- Hu-Friedy, Chicago, IL, USA)

CONTACTS AND LOCATIONS:
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India